CLINICAL TRIAL: NCT07141147
Title: A Prospective, Randomized, Multicenter Clinical Study Comparing Adjuvant Radiotherapy Versus Observation in High-risk Localized Adrenocortical Carcinoma After Surgery.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Chang, vice Director of the Department of Radiation Oncology, Cancer Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-FXY-098
Record Dates: First submitted 2025-08-12; First posted 2025-08-26 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Radiotherapy; High-risk Localized Adrenocortical Carcinoma
Keywords: Adrenocortical carcinoma; Radiotherapy; Multicenter clinical
MeSH Terms: conditions — Adrenocortical Carcinoma | interventions — Radiation

STUDY DESIGN:
Intervention Model Description: This trial uses a simple randomized controlled design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Postoperative Adjuvant Radiotherapy
  Interventions: Radiation: Radiation
- Control group (No Intervention): Regular postoperative follow-up

INTERVENTIONS:
Radiation: Radiation — 1. Technique:Linear accelerator with volumetric modulated arc therapy for irradiation.
  2. Target Volume Delineation (Two-phase irradiation):
  Clinical Target Volume 1 (CTV1):Encompasses tumor bed (preoperative MRI/CT-defined ACC extent) + regional lymphatics (ipsilateral para-aortic nodes).
  Clinical Target Volume 2 (CTV2):Tumor bed only (preoperative MRI/CT-defined ACC extent).
  Planning Target Volume (PTV):PTV1: CTV1 + 0.6 cm margin.PTV2: CTV2 + 0.6 cm margin.
  4.Organs at Risk (OARs):Stomach, liver, bilateral kidneys, pancreas, spinal cord, and bowel/colon within radiation fields.
  5.Prescription Dose: Phase 1: PTV1 → 45 Gy in 25 fractions (1.8 Gy/fraction), 5 fractions/week. Phase 2: PTV2 → 10 Gy in 5 fractions (2.0 Gy/fraction), 5 fractions/week.
  Arms: Experimental group

SUMMARY:
This study is a prospective, randomized, controlled, multicenter clinical trial designed to evaluate whether adjuvant radiotherapy can improve the 3-year recurrence-free survival (RFS) in high-risk localized adrenocortical carcinoma (ACC) patients after radical resection. According to the inclusion and exclusion criteria of the study protocol, 58patients with high-risk localized ACC who underwent radical resection were enrolled and randomly divided into two groups: the control group (Group A), which received regular postoperative follow-up without intervention, and the study group (Group B), which received adjuvant radiotherapy after surgery. The study compared the 3-year RFS and 3-year overall survival (OS) between the two groups and assessed the incidence of grade 3/4 radiotherapy-related adverse reactions, aiming to further clarify the efficacy and safety of postoperative adjuvant radiotherapy.

DETAILED DESCRIPTION:
Adrenocortical Carcinoma (ACC) is an extremely rare and highly aggressive malignant tumor. Its incidence is 0.7-2 per million people, yet it carries a poor prognosis, with an overall 5-year survival rate of only 15-44% . The current standard treatment for localized ACC, defined as European Network for the Study of Adrenal Tumors (ENSAT) stages I-III, is radical surgical resection. However, the postoperative local recurrence rate remains alarmingly high (30-70%) even after complete resection (R0). Therefore, effective adjuvant therapy is crucial for preventing disease recurrence and improving patient survival .

Postoperative adjuvant therapies for ACC include pharmacotherapy and local radiotherapy. Retrospective data suggest that adjuvant mitotane therapy can reduce postoperative recurrence rates and prolong survival in localized ACC. However, the prospective ADIUVO clinical trial showed that adjuvant mitotane did not improve recurrence-free survival (RFS) or overall survival (OS) in low-risk ACC patients post-surgery. Furthermore, 19% of patients permanently discontinued mitotane after a median treatment duration of 6 months due to treatment-related toxicity. Prospective studies on mitotane for adjuvant treatment in high-risk ACC (defined as Ki-67 > 10%, positive resection margin R1, ENSAT stage 3 or higher, or high pathological grade) are currently ongoing [6].

Mitotane has a narrow therapeutic window (14-20 mg/L) and frequently causes severe adverse effects, impacting treatment adherence and quality of life. Reports indicate that all patients taking mitotane develop adrenal insufficiency within months, and 45%-100% develop hypothyroidism, necessitating long-term steroid replacement therapy and hormone level monitoring . Additionally, gastrointestinal reactions (61.5%), neurological symptoms (76.9%), abnormal liver function (50%), and severe cognitive impairment (53.8%) such as memory loss, intellectual dullness, and confusion are common . Hence, there is a pressing need to identify other effective adjuvant treatment strategies.

Local recurrence in localized ACC commonly occurs at the tumor bed and regional lymph nodes, with tumor bed recurrence rates reaching 30%-65% . Among patients with lymph node recurrence, 47% involve para-aortic nodes, with 35% specifically located between the abdominal aorta and inferior vena cava (also part of the para-aortic region) . Therefore, adjuvant radiotherapy targeting the tumor bed and regional lymph nodes holds promise for reducing local recurrence after ACC surgery. Recent retrospective studies suggest that adjuvant radiotherapy may also lower postoperative recurrence rates and improve survival in localized ACC.

A propensity-matched cohort study (n=78) by Gharzai et al. from the University of Michigan showed that the 3-year local RFS rates were 59.5% for surgery plus adjuvant radiotherapy versus 34.2% for surgery alone (P = 0.0035), and the 3-year OS rates were 77.7% versus 48.6% (P = 0.002) . Single-center data from Peking Union Medical College Hospital (Zhu Jiawei et al.) also demonstrated that radiotherapy improved the 3-year local RFS from 38.1% to 77% (P < 0.05). A study of 171 patients with non-metastatic ACC indicated that adjuvant radiotherapy reduced the annual risk of death by 40% (P = 0.02) in patients with positive resection margins . These studies support the use of postoperative adjuvant radiotherapy for ACC patients, particularly those with high recurrence risk.

However, some studies suggest that while adjuvant radiotherapy reduces the local recurrence rate (LRR) in localized ACC, it does not improve OS [15, 16]. Meta-analyses have yielded similar results . Some research even indicates no prognostic benefit. Habra et al. from MD Anderson Cancer Center found 5-year LRR rates of 67% for the radiotherapy group versus 53% for the no-radiotherapy group (P = 0.53) in localized ACC . In other words, the role of postoperative adjuvant radiotherapy in ACC remains controversial.

The European Society for Medical Oncology (ESMO) guidelines do not recommend adjuvant radiotherapy for stage 1-2 localized ACC with R0 resection. For R1 or Rx resections, they suggest individualized therapy combining mitotane and radiotherapy . The National Comprehensive Cancer Network (NCCN) guidelines state that adjuvant radiotherapy may be considered for localized ACC with positive margins, Ki-67 > 10%, tumor rupture, large size, or high pathological grade, but acknowledge a lack of prospective evidence .

In summary, whether adjuvant radiotherapy provides benefits for reducing local recurrence or improving survival in localized ACC post-surgery remains inconclusive. Prospective clinical trials are urgently needed to further evaluate the clinical value of adjuvant radiotherapy in the comprehensive treatment of high-risk localized ACC. We propose conducting a prospective, multicenter randomized controlled trial to investigate whether adjuvant radiotherapy can reduce the 3-year LRR in high-risk localized ACC. The findings have the potential to offer patients better long-term tumor control, provide reliable reference data for ACC adjuvant therapy, and ultimately contribute to the revision of ACC treatment guidelines and the optimization of individualized therapy, holding significant clinical and societal value.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years and ≤ 75 years.
* ECOG performance status score ≤ 1, with an expected survival period ≥ 6 months.
* Completion of radical resection for adrenocortical carcinoma (ACC) with curative intent.
* Postoperative pathological diagnosis of adrenocortical carcinoma.
* Pathological stage is localized ACC: ENSAT stage 1-3; where ENSAT stage 3 is defined as any T stage (T1-4) with regional lymph node positivity, or tumor invasion into surrounding tissues/organs or the renal vein/inferior vena cava, but without distant metastasis.
* High-risk factors: Ki-67 index >10%, ENSAT stage 3, positive resection margin, high pathological grade; the presence of any one of these factors qualifies.
* Postoperative imaging review prior to radiotherapy shows no evidence of residual or metastatic disease.

Exclusion Criteria:

* ENSAT Stage 4 adrenocortical carcinoma.
* Performance status: Karnofsky Performance Status (KPS) score ≤ 70 or Zubrod score > 2.
* Prior radiotherapy to the abdomen or pelvis.
* Insufficient function of major organs (heart, lung, liver, kidney, bone marrow hematopoiesis) precluding tolerance to radiotherapy.
* Pregnant or lactating women, and subjects of childbearing potential unwilling to use contraception.
* Patients with psychiatric disorders, history of alcoholism or substance abuse, or those unable to provide informed consent.
* Other conditions deemed by the investigator to make the subject unsuitable for participation in this trial, including but not limited to: severe illnesses requiring immediate intervention (including psychiatric disorders), severely abnormal laboratory results, or other social or familial high-risk factors.
* Patients with other concurrent primary cancers; or patients diagnosed with another primary malignancy within the 5 years prior to the study (except for adequately treated carcinoma in situ of the cervix, or skin cancers such as basal cell carcinoma, squamous cell carcinoma, or non-melanomatous skin cancer).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
3-year local recurrence-free survival | From a definitive pathological diagnosis to a 3-year follow-up
  The percentage of the patients survive without local recurrence after a time period, from pathological diagnosis

SECONDARY OUTCOMES:
The incidence of grade 3/4 toxicities | The whole period of postoperative adjuvant radiotherapy，an average of 6 weeks
  The percentage of the patients undergo any grade 3/4 toxicity during postoperative adjuvant radiotherapy, based on the Common Terminology Criteria for Adverse Events
3-year overall surviva | From a definitive pathological diagnosis to a 3-year follow-up
  The percentage of the patients survive after a time period, from pathological diagnosis
3-year disease-free survival | From a definitive pathological diagnosis to a 3-year follow-up
  The percentage of the patients survive without local recurrence or distant metastasis after a time period, from pathological diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No